CLINICAL TRIAL: NCT01651169
Title: Evaluating the Effect of Methylphenidate on Intracortical Inhibition in Methamphetamine Abusers Comorbid With Attention Deficit Disorder With Hyperactivity(ADHD) in TMS Unit, Neurcognitive Lab, Iranian National Center for Addiction Studies (INCAS), in 2012. A Randomized, Controlled Trial
Brief Title: Methylphenidate on Intracortical Inhibition in Methamphetamine Abusers Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Khazaeipour, M.D., MPH., Tehran University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: 90-04-49-16359
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Paired Transcranial Magnetic Stimulation; Methamphetamine abuse, ADHD, Methylphenidate; We study the effect of Methamphetamine abuse on Intracortical Inhibition, in ADHD patients, treated with Methylphenidate.
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylphenidate tablets (10mg), ADHD (Experimental): Fifteen patients of ADHD
  Interventions: Other: methylphenidate tablets and Inter-stimulus Intervals (ISI)
- methylphenidate tablets, Methamphetamine abusers and ADHD (Experimental): Fifteen patients of ADHD with Methamphetamine abuse for at least 2 years plus
  Interventions: Other: methylphenidate tablets and Inter-stimulus Intervals (ISI)

INTERVENTIONS:
Other: methylphenidate tablets and Inter-stimulus Intervals (ISI) — We administer 2 single doses of methylphenidate tablets (10mg) separated by a week interval. A paired pulse protocols will be performed with ten single (unconditioned test pulse) and ten paired TMS pulses (conditioning and test pulse) in an intermixed randomized order.
  Short interval cortical inhibition is measured with an Inter-stimulus Intervals (ISI) of 3 msec and a stimulator output of 80% RMT for the conditioning stimulus and 1mVT stimulation intensity for the test stimulus. ICF investigation is measured with an ISI of 13 msec), with the condition of an ISI of 50 msec (ISI 50) and both stimuli applied with 1mVT intensity). Long Interval Cortical Inhibition (LICI) is measured with ISIs of 100 msec (ISI 100), 200 msec (ISI 200), and 300 msec (ISI 300); both stimuli with 1mVT intensity
  Arms: methylphenidate tablets (10mg), ADHD
Other: methylphenidate tablets and Inter-stimulus Intervals (ISI) — We administer 2 single doses of methylphenidate tablets (10mg) separated by a week interval. A paired pulse protocols will be performed with ten single (unconditioned test pulse) and ten paired TMS pulses (conditioning and test pulse) in an intermixed randomized order.
  Short interval cortical inhibition is measured with an Inter-stimulus Intervals (ISI) of 3 msec and a stimulator output of 80% RMT for the conditioning stimulus and 1mVT stimulation intensity for the test stimulus. ICF investigation is measured with an ISI of 13 msec), with the condition of an ISI of 50 msec (ISI 50) and both stimuli applied with 1mVT intensity). Long Interval Cortical Inhibition (LICI) is measured with ISIs of 100 msec (ISI 100), 200 msec (ISI 200), and 300 msec (ISI 300); both stimuli with 1mVT intensity.
  Arms: methylphenidate tablets, Methamphetamine abusers and ADHD

SUMMARY:
Previous studies using transcranial magnetic stimulation (TMS) with paired pulse protocols have shown that a conditioning TMS pulse applied to the human motor cortex changes the excitability of motor pathways from the motor cortex to spinal motorneurons. These effects depended on the stimulus intensity of both conditioning and test pulse and also the ISI). A characteristical sequence of inhibition (short interval cortical inhibition [SICI], GABA-Aerg), facilitation (intracortical facilitation [ICF]), and inhibition again (long interval cortical inhibition [LICI], GABA-Berg) is thought to be physiologically involved in motor control. Previous studies have also shown that neuronal inhibitory motor circuits are also disturbed in ADHD which will be restored by using methylphenidate. In this study the investigators sought to investigate if methamphetamine abuse (from the same chemical class of medications) will alter such effects of methylphenidate.

DETAILED DESCRIPTION:
Design:

Prospective, randomized, -controlled (1:1 randomization), duration-2 single sessions one week apart

Setting:

University psychiatric hospitals in Tehran including Roozbeh Hospital, Rasool Hospital and Imam Hossein General Hospital will refer clients to Iranian National Center for Addiction Studies, Tehran University of Medical Sciences.

Patients:

Fifteen patients with Methamphetamine abuse for at least 2 years plus ADHD are compared with a control group of 15 ADHD patients matched for age and gender

INTERVENTION:

We administer 2 single doses of methylphenidate tablets (10mg) separated by a week interval. A paired pulse protocols will be performed with ten single (unconditioned test pulse) and ten paired TMS pulses (conditioning and test pulse) in an intermixed randomized order.

Short interval cortical inhibition is measured with an Inter-stimulus Intervals (ISI) of 3 msec and a stimulator output of 80% RMT for the conditioning stimulus and 1mVT stimulation intensity for the test stimulus. ICF investigation is measured with an ISI of 13 msec), with the condition of an ISI of 50 msec (ISI 50) and both stimuli applied with 1mVT intensity). Long Interval Cortical Inhibition (LICI) is measured with ISIs of 100 msec (ISI 100), 200 msec (ISI 200), and 300 msec (ISI 300); both stimuli with 1mVT intensity.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Methamphetamine abuse co morbid with ADHD
* Right handedness

Exclusion Criteria:

* Other current Axis I disorders (except simple phobia and nicotine addiction)
* Personal or close family history of seizure disorder
* Ferromagnetic material in body or close to head
* Neurologic disorder
* Pregnancy
* Taking medications known to lower seizure threshold (eg, theophylline)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-11 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Conners ADHD Rating Scale | 1 week
  The primary outcome measure for the study is Conners which measure clinical improvement on ADHD symptoms

SECONDARY OUTCOMES:
Change of Motor Evoked Potential (MEP) | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Javad Alaghband-rad, Tehran University of Medical Sciences, Tehran Province, Iran